CLINICAL TRIAL: NCT01902251
Title: A Phase I, Open-label, Randomized, Parallel, Relative Bioavailability Study Comparing a Capsule and a Tablet Formulation of Enzalutamide Following Multiple Once Daily Doses of 160 mg Enzalutamide in Male Subjects With Prostate Cancer
Brief Title: Relative Bioavailability Study of Enzalutamide in Prostate Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Europe B.V. (Industry)
Collaborators: Medivation, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 9785-CL-0003
Record Dates: First submitted 2013-07-15; First posted 2013-07-18 (Estimated); Last update posted 2014-09-09 (Estimated); Status verified 2014-09

CONDITIONS: Prostate Cancer; Pharmacokinetics of Enzalutamide
Keywords: Phase 1; Prostate cancer; Bioavailability; Food effect; Pharmacokinetics; Xtandi; Enzalutamide; MDV3100
MeSH Terms: conditions — Prostatic Neoplasms | interventions — enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Enzalutamide tablet (Experimental): Multiple once daily oral doses of enzalutamide formulated as a tablet for approximately 8 weeks
  Interventions: Drug: Enzalutamide tablet
- Enzalutamide capsule (Active Comparator): Multiple once daily oral doses of enzalutamide formulated as liquid-filled soft gelatin capsule for approximately 8 weeks
  Interventions: Drug: Enzalutamide capsule

INTERVENTIONS:
Drug: Enzalutamide tablet — Oral
  Other Names: Xtandi; MDV3100
  Arms: Enzalutamide tablet
Drug: Enzalutamide capsule — Oral
  Other Names: Xtandi; MDV3100
  Arms: Enzalutamide capsule

SUMMARY:
A multiple dose relative bioavailability study in patients with prostate cancer comparing a capsule and a tablet formulation of enzalutamide.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed prostate cancer (all stages) for whom androgen deprivation therapy is indicated (except when indicated in a neoadjuvant/adjuvant setting). Subjects may be on ongoing androgen deprivation therapy with a gonadotropin releasing hormone (GnRH) analogue or orchiectomy (i.e., medical or surgical castration) at study entry.
* Progressive disease by Prostate-specific antigen (PSA) or imaging. Disease progression for study entry is defined as one or more of the following 3 criteria:

  * PSA progression defined by a minimum of 2 rising PSA levels with an interval of ≥1 week between each determination. The PSA value during the pre-investigational period should be ≥2 μg/L (2 ng/mL);
  * Soft tissue disease progression defined by the Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST 1.1) for soft tissue disease
  * Bone disease progression defined by two or more new lesions on bone scan

Exclusion Criteria:

* Treatment with chemotherapy within 4 weeks prior to enrollment (Day 1 visit) or plans to initiate treatment with chemotherapy during the study.
* History of seizure or any condition that may predispose to seizure. Also, history of loss of consciousness, or transient ischemic attack within 12 months prior to enrollment (Day 1 visit).
* Patients who previously received treatment with Enzalutamide.
* Concomitant use of drugs that are potent inducers and/or inhibitors of CYP3A4 and CYP2C8.
* Confirmed CYP2C8 poor metabolizer status based on genotyping analysis.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2012-11; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic profile of Enzalutamide under fasted conditions measured by Cmax (Maximum concentration) | Day1 through Day 56 (12 samples)
  Day 56 (fasted) Cmax under steady state conditions of enzalutamide
Pharmacokinetic profile of Enzalutamide under fasted conditions measured by AUC0-24h (Area under the concentration-time curve 0-24h) | Day1 through Day 56 (12 samples)
  Day 56 (fasted) AUC0-24h under steady state conditions of enzalutamide

SECONDARY OUTCOMES:
Pharmacokinetic profile of Enzalutamide under fasted and fed conditions | Day 1, 8, 29, 55, 56 and 57 (38 samples)
  Measured by: Cmax, tmax (Time to attain Cmax), AUC0-24h, Ctrough (Trough concentration), PTR (Peak-trough ratio), CLss/F (Apparent clearance at steady state)
Pharmacokinetic profile of MDPC0001 alone, MDPC0002 alone and sum of Enzalutamide plus MDPC0002 | Day 8, 29, 55, 56 and 57 (26 samples)
  Measured by: Ctrough, Cmax, tmax, AUC0-24h, Ctrough (24h after dosing), PTR
Evaluation of the safety and tolerability of two oral formulations of Enzalutamide assessed through vital signs, adverse events, electrocardiogram and clinical laboratory assessments | Day 1 through Day 58

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Study Manager, Study Director — Astellas Pharma Europe B.V.
Locations (4):
- United States (4):
  - University of Colorado - Anschutz Medical Campus, Denver, Colorado
  - University of Chicago Medical Center, Chicago, Illinois
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - South Texas Accelerated Research Therapeutics, San Antonio, Texas